CLINICAL TRIAL: NCT03226314
Title: Community Epidemiology and Typology of Third-generation Cephalosporins Resistant Enterobacteriaceae (Prevalence, Resistance Mechanisms and Risk Factors) in Reunion Island
Brief Title: Community Epidemiology and Typology of Third-generation Cephalosporins Resistant Enterobacteriaceae in Reunion Island
Acronym: AB-RUN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/CHU/14
Record Dates: First submitted 2017-03-03; First posted 2017-07-21 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Bacterial Resistance
Keywords: bacterial multi-resitance

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — stools samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stool sampled community patients: community patients entering emergency ward or intensive care unit in Reunion Island university hospital and having the stools sampled for bacterial analysis.
  Interventions: Procedure: stool sample

INTERVENTIONS:
Procedure: stool sample — study will be proposed to all patients entering emergency ward or intensive care unit in Reunion Island university hospital. Upon consent, a stool sample will be taken (either directly on emitted stools or by rectal sampling) and analysed for enterobacteriaceae.

SUMMARY:
In its report dated april 2014, World Health Organization confirms antibiotic resistance dissemination in all parts of the world, in hospitals and in community and worries about a possible comeback to a pre-antibiotic era during the 21st century. For the last 15 years, third-generation cephalosporins resistant enterobacteriaceae (3GCREB) prevalence is continuously increasing. Community 3GCREB prevalence has not been studied whereas several observations made in Reunion Island hospital suggest a diffusion in community. In this situation of world-wide and regional extension of bacterial resistance, the investigator offers to study bacterial resistance to antibiotic in Reunion Island community.

DETAILED DESCRIPTION:
The investigator is focused on E. coli species exhibiting BLSE or metallo-betalactamases production that could be encountered du to the increasing level of migratory flow in Reunion Island.

Fecal sample collection will be used for further investigations on bacterial typology.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* aged over 18 years old
* admitted in emergency ward or intensive care of the university hospital of Reunion Island
* who received the patient information notice and who gave their consent
* who have a stool sample performed in the 48 hours following admission
* who understand and can read French

Exclusion Criteria:

Patients:

* transferred from a short-term, middle-term or long-term stay health facility
* who have a stool sample performed more than 48 hours following admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community patients admitted in emergency ward or in intensive care unit for any condition.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Digestive prevalence rate of 3GCREB | through study completion, an average of 1 day
  estimate of digestive prevalence rate of 3GCREB in participating patients and extrapolation to Reunion Island community population.

CONTACTS AND LOCATIONS:
Overall Officials: Julien JAUBERT, MD, Principal Investigator — CHU La Réunion
Locations (1):
- Chu Reunion Island, Saint-Pierre, Reunion Island, Reunion

IPD SHARING:
Plan to Share IPD: No